CLINICAL TRIAL: NCT03948139
Title: Prospective Randomized Study Comparing Functional Bracing vs. Hip Spica Cast in Pediatric Femur Fractures
Brief Title: Femur Fracture: Functional Bracing vs. Hip Spica Cast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: Pediatric Orthopaedic Society of North America (Other)
Responsible Party: Principal Investigator, Lindsay Andras, Assistant Professor of Orthopaedic Surgery, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHLA-18-00233
Record Dates: First submitted 2019-05-08; First posted 2019-05-13 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-06

CONDITIONS: Pediatric Femur Fracture
Keywords: Pediatric; Fracture; Functional Brace; Hip Spica Cast
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Who Masked: Participant
Masking Description: Subjects and parents are blinded until after consent to the study in which they are randomized into the functional brace group or spica cast group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Functional Bracing Group (Other): In a presented abstract, the functional brace group has been to shown equivalent outcomes to the hip spica cast. Subject will be administered the functional brace without going to the operating room to be put under full anesthesia. Most cases will not require any sedation in this group (in some cases, light sedation may be needed). Brace will be used for up to 8 weeks post-administration, until adequate callous formation is confirmed.
  Interventions: Device: Functional Brace
- Spica Cast Group (Other): If subject is randomized into the hip spica cast group, subject will proceed to the operating room and be given general anesthesia to administer the spica cast. Cast will be used for up to 8 weeks, until adequate callous formation is confirmed.
  Interventions: Device: Hip Spica Cast

INTERVENTIONS:
Device: Functional Brace — The study will generate five standardized sized braces based on measurements from prior scans that will be stocked at each institution and modified by the local orthotist to fit the needs of each patient. This will facilitate expedited care while obtaining the same clinical and radiographic results as the fully customized braces. This idea has the potential to be extrapolated to the wider clinical community, creating a true shift in pediatric orthopaedic clinical practice throughout the country.
  Arms: Functional Bracing Group
Device: Hip Spica Cast — Traditional spica casts, the current standard of care for diaphyseal femoral shaft fractures with minimal shortening in children age 0-5 years old. Although spica cast immobilization is standard of care for femur fractures in young children, caring for a child in a spica cast presents a significant socioeconomic burden on families and the healthcare system. Basic hygiene and transportation for a child in a spica cast requires burdensome adjustments for caretakers, as well as the added expenses of specialized car seats or transportation services. Improper spica cast care can lead to skin complications, additional visits for cast adjustments, or even revision casting in the operating room.
  Arms: Spica Cast Group

SUMMARY:
Spica casting is the current standard of care when treating pediatric diaphyseal femur fractures in the 0-5 year age group. A study conducted by Kramer et al. suggests there are both clinical and financial benefits of functional bracing when compared to spica casting. To this date there have been no prospective trials to evaluate these two treatment options. The investigators plan to conduct a multi-center randomized-control trial that will compare the subjective, objective and financial aspects of functional bracing and spica casting for pediatric femur fractures.

DETAILED DESCRIPTION:
Femur fractures are the most common orthopedic injury for which children are hospitalized in the United States. Traditional spica casts, the current standard of care for diaphyseal femoral shaft fractures with minimal shortening in children age 0-5 years old. Although spica cast immobilization is standard of care for femur fractures in young children, caring for a child in a spica cast presents a significant socioeconomic burden on families and the healthcare system. Basic hygiene and transportation for a child in a spica cast requires burdensome adjustments for caretakers, as well as the added expenses of specialized car seats or transportation services. Improper spica cast care can lead to skin complications, additional visits for cast adjustments, or even revision casting in the operating room.

Functional bracing plays an established role in the non-operative management of other long bone fractures in pediatric patients, and offers numerous advantages, including being lightweight, simple to apply, and conducive to hygienic skin care. A study conducted by Kramer et al. suggests there are both clinical and financial benefits of functional bracing when compared to spica casting for femur fractures, including increased patient/parent satisfaction and better cost effectiveness. To date, there have been no prospective trials to confirm these initial findings.

While previous work by Kramer et al demonstrated the advantages of functional bracing when compared to traditional spica casting, the ability to generalize this to other pediatric practices has been limited due to the challenges of making braces in a timely fashion. The braces utilized by Kramer et al require a carver to create a brace with a foot plate that improves rotational control for femur fractures. The cost of a carver is approximately $125,000, and thus few orthotists have access to this piece of equipment. This limits the ability for many pediatric orthopaedists to incorporate functional bracing into their practice.

To make this treatment option more cost effective and accessible, the investigators propose to generate five standardized sized braces based on measurements from prior scans that will be stocked at each institution and modified by the local orthoptist to fit the needs of each patient. This will facilitate expedited care while obtaining the same clinical and radiographic results as the fully customized braces. This idea has the potential to be extrapolated to the wider clinical community, creating a true shift in pediatric orthopaedic clinical practice throughout the country.

The investigators hypothesize that functional bracing will demonstrate equivalent objective outcomes with respect to leg length, time to union, rate of malunion, number of radiographs, and number of clinic visits. The investigators also hypothesize that functional bracing will demonstrate superior economic costs with respect to operating room cost and work days lost for parents, as well as subjective outcomes with respect to Pediatric Outcome Data Collection Instrument, patient/parent satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 0-5 years with an isolated diaphyseal femur fracture. Parents =18 years of age who are cognitively able to take a survey.

Exclusion Criteria:

* Patients >5 years of age without a diagnosis of an isolated diaphyseal femur fracture or polytrauma and those with medical co-morbidities that may affect fracture healing. Parents <18 year of age and unable to take a survey.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
Changes in Leg Length | Radiographs will be reviewed at the pre-op and clinical follow-ups up to 1 year.
  After treatment, leg length will be measured using clinical radiographs to determine if there are any changes to leg length and determine if there are discrepancies.
Changes in union/rate of malunion | Radiographs will be reviewed at the pre-op and clinical follow-ups up to 1 year.
  This will be measuring the length of time and changes in union of bone, and to see if the bone has not healed properly.
Number of radiographs and clinic visits | This will be reviewed and counted for up to 1 year.
  This will be used to determine which arm had less radiation from radiographs and less visits with the surgeon.
Economic costs (operating room cost) | This will be examined at the 1 day of intervention.
  This will be to compare the economic costs between the administration of a spica cast vs. a functional brace.
Work days lost for parents | This will be surveyed at the 6 week post-intervention visit.
  This will be collected from a parent reported outcome survey which will help determine the amount of days a parent lost to work due to their child's condition.
Work days lost for parents | This will be surveyed at the 1 year post-intervention visit.
  This will be collected from a parent reported outcome survey which will help determine the amount of days a parent lost to work due to their child's condition.
Pediatric Outcome Data Collection Instrument (PODCI) | This will be surveyed at the 6 week post-intervention visit.
  The PODCI is a validated quality of life and outcome questionnaire used for various pediatric orthopaedic studies. It will allow the study team to determine the subjective outcomes of the subject.This will also be completed by the parent.
Pediatric Outcome Data Collection Instrument (PODCI) | This will be surveyed at the 1 year post-intervention visit.
  The PODCI is a validated quality of life and outcome questionnaire used for various pediatric orthopaedic studies. It will allow the study team to determine the subjective outcomes of the subject.This will also be completed by the parent.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Andras, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (2):
- United States (2):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No